CLINICAL TRIAL: NCT02865928
Title: Serratus Plane Block for Postoperative Pain Control After Breast Surgery
Brief Title: Serratus Plane Block for Postoperative Pain Control
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We decided to terminate this study due to staffing changes and other limitations posed by the COVID-19 pandemic.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Judith Aronsohn, MD, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-246
Record Dates: First submitted 2016-06-28; First posted 2016-08-15 (Estimated); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Outpatient Breast Surgery; Mastopexy; Augmentation; Revision
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivicaine HCl (Experimental): Ultrasound guided serratus plane block with bupivacaine HCl.
  Interventions: Drug: Bupivicaine HCl
- Normal Saline (Placebo Comparator): Placebo injection on operated side, same technique as experimental group.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Bupivicaine HCl — Ultrasound guided serratus plane block with bupivicaine
  Other Names: Bupivicaine
  Arms: Bupivicaine HCl
Drug: Normal Saline — Same injection technique as intervention arm with normal saline
  Other Names: 0.09% NaCl
  Arms: Normal Saline

SUMMARY:
This is a randomized, double-blinded, placebo-controlled trial of serratus plane blocks in subjects undergoing outpatient unilateral or bilateral breast surgery. Ninety subjects will be enrolled into the study at presurgical testing. Subjects will be stratified based on surgery type and randomized to receive a serratus plane block with either bupivicaine HCL or placebo. All patients will receive standard intraoperative anesthesia and standard postoperative pain control. The primary endpoint is the amount of opioid administered postoperatively. Secondary endpoints include postoperative pain intensity at timed intervals, amount of opioid administered intraoperatively and postoperatively, incidence of nausea and vomiting, time to discharge and patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III.
* Undergoing outpatient breast surgery requiring general anesthesia, including but not limited to mastectomy, lumpectomy, reconstruction with tissue expanders or implants and reconstruction revision.

Exclusion Criteria:

* Unable to provide informed consent.
* Patients who are pregnant or nursing.
* ASA IV-V.
* Alcohol or narcotic dependence in the last 2 years.
* Concurrent condition requiring regular use of analgesia that may confound post-surgical assessments as determined by principle investigator.
* Hepatic disease.
* Allergies to amide anesthetics as determined from medical history or patient self-report.
* Evidence of infection at injection site.
* Contraindication to pain medications such as acetominophen, morphine, oxycodone, keterolac, dilaudid, Toradol.
* Body weight <50kg.
* BMI>40kg/m2.
* History of hypotension.
* Abnormal renal (creatinine > 1.5 mg/dL) function.
* Heart block.
* Any physical, mental or medical condition, that in the opinion of the investigator, makes study participation inadvisable.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Aronsohn, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health System, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At pre-surgical testing, approximately one week before surgery, potential subjects will be screened and recruited into the trial.
Pre-assignment Details: * Any physical, mental or medical condition, makes study participation inadvisable. For example, chronic pain conditions, significant medical disease, laboratory abnormalities or condition(s) that could impact a subject's ability to communicate with the study staff, complete study activities such as provide pain scores, or would otherwise contradict study participation
  * Patients who are pregnant or nursing.
  * Patients may withdraw from this study at their discretion.
Period: Overall Study
Arm/Group | Bupivicaine HCl | Normal Saline
Started | 22 | 20
Completed | 19 | 19
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Subject is a screen failure. Miscommunication with the randomization request. | 1 | 0
Not completed — Patient experience and satisfaction category lost one patient in each group to follow-up call. | 1 | 1

BASELINE CHARACTERISTICS:
Population: At pre-surgical testing, subjects screened will be recruited into the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivicaine HCl | Normal Saline | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Full Range); unit: years] | 52.045 [23 to 70] | 49.05 [30 to 65] | 50.62 [23 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 18 | 14 | 32
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 16 | 12 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Requirements
Description: Postoperatively, oral and IV rescue medication will be administered to both groups upon request as per standard of care. The use of narcotics will also be recorded intra-operatively, for the duration of PACU and hospital stay and up until the end of postoperative day one. Consumption of rescue medication will be converted to the morphine equivalent (ME) dose for analysis.
Time Frame: 4 to 10 hours
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Groups:
- Bupivacaine HCl: Ultrasound guided serratus plane block with bupivacaine HCl.
  Bupivicaine HCl: Ultrasound guided serratus plane block with bupivicaine
Arm/Group | Bupivacaine HCl | Normal Saline
Number analyzed (Participants) | 22 | 20
Morphine Milligram Equivalents (MME) | 19.875 (21.93703609496) | 17.5 (22.124052165246)

2. Secondary Outcome: Postoperative Pain With Numeric Rating Scale
Description: * Postoperatively, pain intensities at rest and on movement will be assessed every 30 minutes in the PACU for the first four hours and at hourly intervals up until PACU discharge, using the visual analog scale (VAS) with two anchor points; 0 being no pain and 10 being the worst pain imaginable. Pain scores were combined to find the mean and standard deviation.
  * The study will collect pain and scores in the PACU every 30 minutes up to 4 hrs and at 1 hr intervals after 4 hours for the duration of PACU stay.
Time Frame: every 30 minutes in the PACU for the first four hours and at hourly intervals up until PACU discharge, up to 10 hours.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine HCl | Normal Saline
Number analyzed (Participants) | 22 | 20
score on a scale | 0.7818181818181 (0.8138642058897) | 0.7536363636363 (0.7338097362481)

3. Secondary Outcome: Postoperative Nausea and Vomiting With Verbal Rating Scale
Description: Nausea assessed at time intervals with numeric rating scale and episodes of vomiting and retching recorded.
  * Evaluation will be performed at every 30 minutes in the PACU for the first four hours and at hourly intervals up until PACU discharge using a standard 11-point verbal rating scale, for which "0" represents "no nausea" and 10 represents "worst nausea imaginable." Nausea and vomiting scores were combined to find the mean and standard deviation.
  * The study will collect nausea and scores in the PACU every 30 minutes up to 4 hrs and at 1 hr intervals after 4 hours for the duration of PACU stay.
Time Frame: every 30 minutes in the PACU for the first four hours and at hourly intervals up until PACU discharge, up to 10 hours.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine HCl | Normal Saline
Number analyzed (Participants) | 22 | 20
score on a scale | 0.2545454545454 (0.4842899494217) | 0.3363636363636 (0.8099533063187)

4. Secondary Outcome: Number of Participants Who Required Antiemetics During the Postoperative Period.
Description: Number of Participants who Required Antiemetics During the Postoperative Period.
Time Frame: 4 to 10 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine HCl | Normal Saline
Number analyzed (Participants) | 22 | 20
Participants | 6 | 5

5. Secondary Outcome: PACU Length of Stay
Description: Time to PACU discharge
Time Frame: 0 to 10 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Bupivacaine HCl | Normal Saline
Number analyzed (Participants) | 22 | 20
Minutes | 115.8 (48.879658884157) | 144.35 (83.998292589163)

6. Secondary Outcome: Patient Experience and Satisfaction With a 5-point Categorial Scale
Description: This survey assessed patient experience and satisfaction. The scale ranged from "Very dissatisfied" or "1" was the minimum value. "Very satisfied" or "5" was the maximum value.
Time Frame: 1 week
Population: One patient in each group (Bupivacaine HCI & Normal Saline) was missing information on patient satisfaction with pain management.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine HCl | Normal Saline
Number analyzed (Participants) | 19 | 19
score on a scale
  Anesthesia Satisfaction | 4.4210526315789 (0.6069769786668) | 4 (1.0540925533894)
  Surgery Satisfaction | 4.2631578947368 (0.9911892555667) | 4.2105263157894 (0.6306035352846)

ADVERSE EVENTS:
Time Frame: The protocol states that all adverse events occurring during the study period will be recorded. The clinical course of each event will be followed until resolution, stabilization, or until it has been determined that the study treatment or participation is not the cause. This will occur through study completion, an average of 1 year.
Description: The investigator will seek information on AE by monitoring while subject is under anesthesia, specific questioning and by examination. All related signs, symptoms, and abnormal diagnostic procedures results will be recorded in the source document. All AEs occurring during the study period will be recorded. The clinical course of each event will be followed until resolution, stabilization, or until it has been determined that the study treatment or participation is not the cause
Arm/Group | Bupivicaine HCl | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT02865928/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT02865928/ICF_001.pdf